CLINICAL TRIAL: NCT05873322
Title: Glucose Intolerance and Diabetes Related to Treatment With Steroids and PEG- Asparaginase in Children and Adolescents With ALL and Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, MD, PhD, Associate Professor, Aarhus University Hospital
Other Study IDs: Glucose intolerance
Record Dates: First submitted 2023-01-25; First posted 2023-05-24 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Drug-Induced Diabetes Mellitus; Impaired Glucose Tolerance; Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Glucose Intolerance; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall survival of acute lymphoblastic leukemia (ALL) and lymphoma in children and adolescents is above 90%. The survival rate has increased significantly during the last decades as a consequence of more intensive chemotherapy. This very toxic treatment results in severe acute toxicities and late effects, which is the biggest challenge today besides survival. The overall purpose of contemporary ALL treatment is to reduce the toxic treatment without compromising the excellent survival rates of these diseases. This study is a part of this. The researchers want to investigate the incidence of glucose intolerance and medicine induced diabetes during treatment for ALL and lymphoma with steroids (prednisolone or dexamethasone) and ± PEG-asparaginase.

Steroids and asparaginase are used in the treatment of ALL and lymphomas, and both drugs may induce glucose intolerance or diabetes, especially when they are given concomitantly. The incidence and duration of increased blood glucose levels are not very well investigated, and especially not monitored continuously during treatment phases with steroids and +/- asparaginase, as the investigators want to do in this study.

In the study the participants must have a glucose sensor attached under the skin, which continuously measures blood glucose during treatment. Moreover, blood samples are drawn several times to measure insulin sensitivity and beta cell function.

The participants are children and adolescents (1.0-17.9 years) with newly diagnosed ALL or lymphoma treated at one of the four Danish pediatric oncology sites.

Blood glucose levels are followed during treatment with steroids and PEG-asparaginase in these patient groups. The results may give rise to a new treatment guidelines for measuring and treating blood glucose in these patients. In the future this may help reduce the development of type 2 diabetes mellitus and metabolic syndrome in survivors of ALL and lymphoma.

DETAILED DESCRIPTION:
Purpose:

Survival rates for acute lymphoblastic leukemia (ALL) have improved during the last decades. Accordingly, the research now also focuses more on reducing the acute toxicities during treatment and the risk of late effects after treatment without compromising overall survival.

Main aim:

To investigate the incidence and severity of medication induced glucose intolerance and diabetes mellitus in children and adolescents (1.0-17.9) treated for acute lymphoblastic leukemia or lymphoma.

Secondary aim:

To translate the results of the project to new treatment guidelines in relation to measuring and treating glucose level during treatment

Background:

ALL is the most common malignant disease in childhood. The overall survival after ALL has increased significantly during the last decades, and is now above 90% on most contemporary treatment protocols. Due to very toxic treatment with chemotherapy more than 50% of the patients experience severe acute toxicities, and severe late effects that influence daily life and quality of life are expected in approximately 50% of the patients.

Lymphomas (Hodgkin and non-Hodgkin, HL and NHL) are rare diseases in childhood, but the incidence increases in adolescence. The prognosis is good (>90%).

Children and adolescents with ALL and lymphoma are treated with steroids (dexamethasone or prednisolone) and +/- the enzyme PEG-Asparaginase (PEG-Asp).

During treatment some of the patients develop medication induced glucose intolerance with blood glucose levels (BG) after a meal between 7-11 mmol/l, and some develop diabetes mellitus (DM) with fasting BG >7 mmol/l or BG after a meal >11 mmol/l. Hyperglycemia during ALL induction (first part of the treatment) is associated with a poorer prognosis.

Dexamethasone and to a lesser extent prednisolone may induce an insulin resistant state, while asparaginase may cause pancreatitis including beta cell dysfunction, with reduced insulin secretion and subsequently DM. The incidence and severity of these medication induced blood glucose changes are very limited investigated in children and adolescents with ALL and lymphoma.

Our knowledge of glucose intolerance and medication induced diabetes in this group of patients is primarily based on retrospective studies. Data on continuous glucose monitoring in these patient groups have not been published earlier.

Combination of steroids and asparaginase treatment induces hyperglycemia in 10 to 20% of the patients. In the current Western European ALL protocol (ALLTogether), in which the Nordic Countries participate anthracyclines are omitted for more than 50% of the patient for the prevention of cardiac late effects, and instead the treatment of asparaginase is advanced compared to previous Nordic/Baltic treatment protocols and thus given concomitant with steroids, like in some lymphoma protocols. Knowledge of the influence of this on the glucose metabolism and possible late effects is lacking.

It has been shown, that age >10 years and overweight are risk factors for development of medication-induced diabetes. Approximately 80% of the ALL-cohort is <10 years of age, while most lymphoma patients are ≥ 10 years. By including both ALL and lymphoma patients, it will be possible to compare both types of steroids, steroid ±PEG-Asp and age.

The high cure rate has a cost. Treatment related severe acute toxicities are common. Invasive infections are among the most common acute side effects to the toxic treatment. Hyperglycemia, especially during induction therapy, has been shown to increase the risk for neutropenic fever and invasive fungal infections as well as the severity of the infections leading to increased hospitalization and potentially increased treatment related mortality.

Metabolic syndrome is among the most frequent reported late effects after ALL. There seems to be an increased risk of metabolic syndrome in ALL patients who have suffered from medication-induced diabetes.

Medication induced diabetes while receiving treatment for ALL also seems to cause an increased risk for prediabetes and type 2 diabetes mellitus (T2DM) in adult survivors after ALL in childhood.

Hypothesis:

* 10% of the patients in combination treatment with dexamethasone and PEG- asparaginase will develop DM
* 15-20% of the patients in combination treatment will develop glucose intolerance for 50% of the time
* 2-5% of the patients who receive monotherapy with either dexamethasone or prednisolone will develop DM
* 10-15% of the patients who receive monotherapy with either dexamethasone or prednisolone will develop glucose intolerance for 50% of the time.

The majority of cases are expected to be above 10 years.

Methods:

The study is a prospective study, where the investigators by continuous glucose monitoring (CGM) investigate the patients' blood glucose profiles during treatment with steroids (dexamethasone/prednisolone) and ± PEG-asparaginase (monotherapy or combination treatment).

The participants must have a glucose sensor attached under the skin, which continuously measures blood glucose during treatment. The glucose sensor is inserted using a thin needle inside a so-called applicator. The blood glucose measurements are blinded to the patient and the treating team. Moreover, blood samples are drawn several times to measure insulin sensitivity and beta cell function.

The researchers want:

1. To do BG profiles by CGM in ALL and lymphoma patients in order to estimate the incidence of medication induced glucose intolerance and DM in different age groups (</>=10 years), different steroids (dexa/pred), and ± in combination with PEG-Asp.
2. To measure the duration of BG >10 mmol/l in the patients during treatment.
3. To describe the extent of insulin sensitivity and beta cell function before, during and after treatment.
4. To measure the duration of the changes in insulin sensitivity and the beta cell function.
5. To describe the association between the BG-profiles and the asparaginase enzyme activity levels.

Study blood tests will be planned in parallel with other visits at the hospital according to treatment protocol.

Study population:

The study population will consist of:

* All children and adolescents (1.0-17.9 years) with newly diagnosed ALL and treated according to the current protocol at one of the four Danish Pediatric sites.
* All children and adolescents (1.0-17.9 years) with newly diagnosed HL or NHL at one of the four Danish Pediatric sites.

In Denmark 40 new cases aged 1.0-17.9 years are diagnosed yearly with ALL and 18 with lymphoma. It is expected that approximately 75% will consent to the study, leaving inclusion of 44 patients annually. The aim is to include at least 100 patients during three years.

Investigations:

The Dexcom G6 device for CGM is reliable with exact BG measurement at low BG levels as well at high BG levels, and it is the device that will be used for CGM. It has to be changed every 10th day. Data is transferred wireless by a data transmitter to a receiver and blinded to the patient and treating team. Appointed persons from the study group will have access to the data in order to make sure that the devices and transferal of data is working satisfactory.

Other investigations:

1. Just before steroid induction therapy, blood samples are drawn for HbA1c, fasting BG, insulin, C-peptide as well as DM specific autoantibodies (GAD-65, IA2 A, Zink AB) in order to evaluate insulin sensitivity and beta cell function.
2. Application of Dexcom for CGM until at least 10 days after termination of steroid ± PEG-Asp treatment (including tapering).
3. Blood samples for measurement of HbA1c, fasting BG, insulin, C-peptide, pancreas-specific amylase and lipase at specific time points depending on diagnosis and treatment phase. A blood sample for measurement of DM specific autoantibodies is drawn after therapy termination.
4. Levels of asparaginase enzyme activity will be included in treatment phases, where asparaginase is given concomitant to steroids. The measurements are done as standard of care in the A2G-protocol.

The study follow-up (i.e., visits for renewal of the Dexcom sensor and the transmitter as well as the blood tests) is quite extensive, why in order to ensure all data, affiliation of dedicated research nurses at the four departments are required.

Statistics and sample size determination:

Comparisons of repeated measurements over time of blood sugars during treatment with steroids, dexamethasone and prednisolone, and with and without concomitant asparaginase treatment will be done using linear mixed models. If the measurements are not normally distributed, they will be transformed in order to achieve a normal distribution. The regression models will be adjusted for relevant parameters such as age and gender. Two-way interactions between covariates will be tested.

Generalized linear mixed models will be used for comparison of patients with glucose intolerance and DM on mono therapy and combination therapy, respectively.

Perspectives:

The results of the study may give rise to new monitoring and treatment guidelines for glucose intolerance and medicine-induced diabetes during treatment for ALL and lymphoma. A follow-up study in 5 or 10 years will be able to elucidate the importance of hyperglycemia for the development of T2DM, metabolic syndrome (or precursor to this). This will contribute to better treatment and follow up as prolonged hyperglycemia is associated with increased risk of infections during treatment, possible decreased survival after ALL and T2DM or metabolic syndrome later in life.

In the present Western European ALL treatment protocol (ALLTogether1), dexamethasone and PEG-asparaginase is given in combination. This is not very well investigated, and in particular data on continuous glucose monitoring as well as data on the association between BG and enzyme activity levels have not been published earlier.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents diagnosed with ALL and Lymphoma and treated according to the established and approved treatment protocols for these diseases in Denmark can be included in the study.

Exclusion Criteria:

* Children and adolescents not fulfilling the inclusion criteria.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: All children and adolescents (1.0-17.9 years) with newly diagnosed ALL or lymphoma and treated in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related impaired glucose tolerance | CGM is used from the beginning of ALL/lymphoma treatment day 1 and in up to 120 days. For the ALL patient in the induction phase, consolidation 2 and delayed intensification phase
  Glucose levels are measured using the technology continuous glucose monitoring (CGM). A glucose sensor is attached under the skin which continuously measures the glucose level every 5 minutes during treatment with steroids or PEG-Asparaginase. Impaired glucose tolerance is defined as a blood glucose (BG) 2 hours after a meal between 7.8-11 mmol/l
Number of participants with treatment-related diabetes | CGM is used from the beginning of ALL/lymphoma treatment day 1 and in up to 120 days. For the ALL patient in the induction phase, consolidation 2 and delayed intensification phase
  Glucose levels are measured using the technology continuous glucose monitoring (CGM). A glucose sensor is attached under the skin which continuously measures the glucose level every 5 minutes during treatment with steroids or PEG-Asparaginase. Diabetes is defined as a fasting BG ≥7 mmol/l or BG after a meal ≥ 11.1 mmol/l.
The extent of insulin resistance at baseline | Fasting plasma glucose and insulin are measured at baseline
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 5 | Fasting plasma glucose and insulin are measured at week 5
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 8 | Fasting plasma glucose and insulin are measured at week 8
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 12/13 | Fasting plasma glucose and insulin are measured at week 12/13. Which week depends on which risk group the patient belongs to.
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 15/16 | Fasting plasma glucose and insulin are measured at week 15/16. Which week depends on which risk group the patient belongs to.
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 18/19 | Fasting plasma glucose and insulin are measured at week 18/19. Which week depends on which risk group the patient belongs to.
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 20/21/22 | Fasting plasma glucose and insulin are measured at week 20/21/22. Which week depends on which risk group the patient belongs to.
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of insulin resistance at week 22/23/28 | Fasting plasma glucose and insulin are measured at week 22/23/28. Which week depends on which risk group the patient belongs to.
  Insulin resistance is calculated from the homeostasis model assessment of insulin resistance using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at baseline | Fasting plasma glucose and insulin are measured at baseline
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 5 | Fasting plasma glucose and insulin are measured at week 5.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 8 | Fasting plasma glucose and insulin are measured at week 8.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 12/13 | Fasting plasma glucose and insulin are measured at week 12/13. Which week depends on which risk group the patient belongs to.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 15/16 | Fasting plasma glucose and insulin are measured at week 15/16. Which week depends on which risk group the patient belongs to.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 18/19 | Fasting plasma glucose and insulin are measured at week 18/19. Which week depends on which risk group the patient belongs to.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 20/21/22 | Fasting plasma glucose and insulin are measured at week 20/21/22. Which week depends on which risk group the patient belongs to.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin
The extent of beta cell function at week 22/23/28 | Fasting plasma glucose and insulin are measured at week 22/23/28. Which week depends on which risk group the patient belongs to.
  Beta cell function is calculated from the homeostasis model assessment of beta cell function using fasting plasma glucose and fasting plasma insulin

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark